CLINICAL TRIAL: NCT04869267
Title: Effectiveness of Acceptance and Commitment Therapy on Fatigue Interference and Health-related Quality of Life Among Patients With Advanced Lung Cancer: A Randomized Controlled Trial
Brief Title: Acceptance and Commitment Therapy in Patients With Advanced Lung Cancer
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Huiyuan LI, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CREC Ref. No. 2020.581
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer; Advanced Cancer
Keywords: lung cancer; palliative care; Acceptance and Commitment Therapy; fatigue; health-related quality of life
MeSH Terms: conditions — Lung Neoplasms; Fatigue | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study. Participants in Group A receive Acceptance and Commitment Therapy based on usual care. Participants in Group B receive usual care.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors who are independent with the research will be trained before formally conducting data collecting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT group (Experimental): Participants in the intervention group will receive ACT intervention, consisting of four individual sessions (First session by face to face, the last three sessions by Wechat) of 60-90 min each (once/week), in addition to usual care.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Usual care group (Other): Participants randomized to the control group will receive usual care, including treatments and daily care during admission, medication instructions, diet and exercise advice, retest recommendations when discharge.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Session 1:
  This session aims to let the participants get familiar with the interventionist. The interventionist will tell them the purpose of the program and basic rules. And the interventionist will promise their privacy protection.
  Session 2:
  This session includes how to separate thoughts/feelings/sensations related to diagnose with advanced lung cancer and experience of fatigue with facts and see these feelings in an objective way with observing self.
  Session 3:
  This session mainly aims to help participants understand the importance of values, differentiate values from goals and clarify their personal values.
  Session 4:
  This session aims at helping patients practice to engaging in committed action based on chosen values, motivated to change behavior in consistency with life direction and health goal.
  Arms: ACT group
Other: Usual care — The usual care mainly includes treatments and daily care during admission, medication instructions, diet and exercise advice, retest recommendations when discharge
  Arms: Usual care group

SUMMARY:
Lung cancer is a malignant tumor that has transformed from a single cancer disease into one of the most striking global health problems. Lung cancer has an insidious onset, and most patients are first diagnosed with the middle and advanced stage. Cancer related fatigue is the most common and distressing symptom reported by lung cancer patients. For cancer patients, fatigue has lasting impact on physical, psychological and social functions, interferes with activities and participating in life events, thereby worsening the health-related quality of life. Acceptance and Commitment Therapy (ACT) is the third-wave cognitive behavioral therapy to improve functioning and health-related quality of life by increasing psychological flexibility. The study aims to examine the effectiveness of ACT on fatigue interference and health-related quality of life in patients with advanced lung cancer.

DETAILED DESCRIPTION:
A two-arm, assessor-blind randomized controlled trial will be conducted to investigate the effects of ACT on advanced lung cancer patients compared to usual care. Participants in the same ward will be randomized at a 1:1 ratio to the intervention group or control group. Block randomization will be conducted by an independent research assistant using randomly varying block size of 4, 6 to avoid selection bias. The study aims to examine the effectiveness of ACT on fatigue interference and health-related quality of life in patients with advanced lung cancer. The Specific objectives are: 1) To investigate the effects of ACT on primary outcomes: fatigue interference and health-related quality of life compared to control group at post-intervention and three months follow-up. 2) To investigate the effects of ACT on the secondary outcomes: cancer-related fatigue, depressive symptoms, anxiety, distress and exercise capacity and process outcomes including psychological flexibility, ACT related variables (acceptance and cognitive defusion) at post-intervention and three months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 or over;
2. diagnosed with stage III or stage IV lung cancer by pathological section or cytology;
3. experienced unexplained fatigue syndrome: the score of 3 or more on the Fatigue Symptom Inventory (FSI); and
4. able to provide informed consent and effectively collect data.

Exclusion Criteria:

1. diagnosed with cognitive dysfunction or other mental illnesses that may interfere with their completion of treatment;
2. who are with a life expectancy <3 months, or whose physical conditions are considered ineligible for the present study based on the physician's judgment; and
3. who are receiving or have just completed other lung cancer-related intervention programs within the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the score of fatigue interference assessed by The Fatigue Symptom Inventory at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 4-week intervention)
  A 13-item instrument that measures the intensity and interference of fatigue over the previous 7 days. The first four items are used to assess the intensity of fatigue, Item 5 - Item 11 are to assess the degree to which fatigue in the past week was judged to interfere with different aspects, such as general activity, bathe and dress ability, work activity, concentration ability, relation with others, enjoyment of life and mood, using a 11-point Likert scale ranging from 0 (no interference) to 10 (extreme interference). 0 indicates no fatigue and 127 indicates the worst fatigue intensity and interference.
  Change= (One week after the intervention score - Baseline score)
Change from baseline in the score of the score of fatigue interference assessed by The Fatigue Symptom Inventory at three months after the 4-week intervention | Baseline (T0) and three months follow-up (T2, three months after the 4-week intervention)
  A 13-item instrument that measures the intensity and interference of fatigue over the previous 7 days. The first four items are used to assess the intensity of fatigue, Item 5 - Item 11 are to assess the degree to which fatigue in the past week was judged to interfere with different aspects, such as general activity, bathe and dress ability, work activity, concentration ability, relation with others, enjoyment of life and mood, using a 11-point Likert scale ranging from 0 (no interference) to 10 (extreme interference). 0 indicates no fatigue and 127 indicates the worst fatigue intensity and interference.
  Change= (Three months after the intervention score - Baseline score)
Change from baseline in the score of health-related quality of life assessed by Functional Assessment of Cancer Therapy - Lung, Version 4 at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 4-week intervention)
  36 items scored from 0 (not at all) to 4 (very much) to assess QoL of lung cancer patients, including 5 domains: physical, social/family, emotional, and functional well-being, and additional concerns about lung cancer. The overall score can be obtained by adding all subscale scores. 0 indicates no quality of life and 144 indicates the highest quality of life.
  Change= (One week after the intervention score - Baseline score)
Change from baseline in the score of health-related quality of life assessed by Functional Assessment of Cancer Therapy - Lung, Version 4 at three months after the 4-week intervention | Baseline (T0) and three months follow-up (T2, three months after the 4-week intervention)
  36 items scored from 0 (not at all) to 4 (very much) to assess QoL of lung cancer patients, including 5 domains: physical, social/family, emotional, and functional well-being, and additional concerns about lung cancer. The overall score can be obtained by adding all subscale scores. 0 indicates no quality of life and 144 indicates the highest quality of life.
  Change= (Three months after the intervention score - Baseline score)

SECONDARY OUTCOMES:
Change from baseline in the score of cancer related fatigue assessed by The Multidimensional Fatigue Inventory at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 4-week intervention)
  20-item self-reported instrument testing the subjective experience of fatigue. 20 indicates the low level of fatigue and 80 indicates the high level of fatigue. 20 indicates low level of fatigue and 80 indicates the high level of fatigue.
  Change= (One week after the intervention score - Baseline score)
Change from baseline in the score of cancer related fatigue assessed by The Multidimensional Fatigue Inventory at three months after the intervention | Baseline (T0) and three months follow-up (T2, three months after the 4-week intervention)
  20-item self-reported instrument testing the subjective experience of fatigue. 20 indicates the low level of fatigue and 80 indicates the high level of fatigue. 20 indicates low level of fatigue and 80 indicates the high level of fatigue.
  Change= (Three months after the intervention score - Baseline score)
Change from baseline in the score of depressive symptoms assessed by The Patient Health Questionnaire (PHQ-9) at one week after the intervention. | Baseline (T0) and post-intervention (T1, one week after the 4-week intervention)
  A 9-item scale to measure the severity of depressive symptom ranged from 0 to 27, in which each item can be score from 0 (not at all) to 3 (nearly every day). 0 indicates no depression and 27 indicates severe depression.
  Change= (One week after the intervention score - Baseline score)
Change from baseline in the score of depressive symptoms assessed by The Patient Health Questionnaire (PHQ-9) at three months after the intervention. | Baseline (T0) and three months follow-up (T2, three months after the 4-week intervention)
  A 9-item scale to measure the severity of depressive symptom ranged from 0 to 27, in which each item can be score from 0 (not at all) to 3 (nearly every day). 0 indicates no depression and 27 indicates severe depression.
  Change= (Three months after the intervention score - Baseline score)
Change from baseline in the score of anxiety assessed by Generalized Anxiety Disorder Scale (GAD-7) at one week after the intervention. | Baseline (T0) and post-intervention (T1, one week after the 4-week intervention)
  A brief self-report instrument to measure severity of anxiety with 7 items ranged from 0 to 21. 0 indicates no anxiety and 21 indicates severe anxiety.
  Change= (One week after the intervention score - Baseline score)
Change from baseline in the score of anxiety assessed by Generalized Anxiety Disorder Scale (GAD-7) at three months after the intervention. | Baseline (T0) and three months follow-up (T2, three months after the 4-week intervention)
  A brief self-report instrument to measure severity of anxiety with 7 items ranged from 0 to 21. 0 indicates no anxiety and 21 indicates severe anxiety.
  Change= (Three months after the intervention score - Baseline score)
Change from baseline in the score of psychological distress assessed by Impact of Events Scale -Revised version at one week after the intervention. | Baseline (T0) and post-intervention (T1, one week after the 4-week intervention)
  It has 22 items containing three domains: Intrusion, Avoidance, and Hyperarousal subscales using a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely) ranged from 0 to 88. 0 indicates low level of distress and 88 indicates severe distress.
  Change= (One week after the intervention score - Baseline score)
Change from baseline in the score of psychological distress assessed by Impact of Events Scale -Revised version at three months after the intervention. | Baseline (T0) and three months follow-up (T2, three months after the 4-week intervention)
  It has 22 items containing three domains: Intrusion, Avoidance, and Hyperarousal subscales using a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely) ranged from 0 to 88. 0 indicates low level of distress and 88 indicates severe distress.
  Change= (Three months after the intervention score - Baseline score)
Change from baseline in exercise capacity assessed by self-designed questions at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 4-week intervention)
  Including the type of exercise (What kind of exercise do you usually do?); the intensity of exercise (What intensity of exercise do you usually do? Low/moderate/high?); frequency of exercise per week (How many times do you exercise on average a week?); and the duration of exercise each time (min) (How long will you take each exercise?) Change= (One week after the intervention score - Baseline score)
Change from baseline in exercise capacity assessed by self-designed questions at three months after the intervention | Baseline (T0) and three months follow-up (T2, three months after the 4-week intervention)
  Including the type of exercise (What kind of exercise do you usually do?); the intensity of exercise (What intensity of exercise do you usually do? Low/moderate/high?); frequency of exercise per week (How many times do you exercise on average a week?); and the duration of exercise each time (min) (How long will you take each exercise?) Change= (Three months after the intervention score - Baseline score)
Change from baseline in the score of psychological flexibility assessed by Comprehensive assessment of Acceptance and Commitment Therapy processes at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 4-week intervention)
  A comprehensive ACT process measure to evaluate the level of psychological flexibility (and constituent sub-process) within the ACT model with 18 items ranged from 18 to 90. 18 indicates low level of psychological flexibility and 90 indicates the high level of psychological flexibility.
  Change= (One week after the intervention score - Baseline score)
Change from baseline in the score of psychological flexibility assessed by Comprehensive assessment of Acceptance and Commitment Therapy processes at three months after the intervention | Baseline (T0) and three months follow-up (T2, three months after the 4-week intervention)
  A comprehensive ACT process measure to evaluate the level of psychological flexibility (and constituent sub-process) within the ACT model with 18 items ranged from 18 to 90. 18 indicates low level of psychological flexibility and 90 indicates the high level of psychological flexibility.
  Change= (Three months after the intervention score - Baseline score)
Change from baseline in the score of acceptance assessed by Acceptance and Action Cancer Questionnaire at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 4-week intervention)
  18-item questionnaire to measure experiential avoidance, in which participants response the possibility that they accept or avoid repulsive thoughts and feelings to each item using a 7-point Likert scale (1 = never true to 7 = always true) ranged from 18 to 126. The higher the overall score, the greater level of experiential avoidance or low level of acceptance. 18 indicates low level of acceptance and 90 indicates the high level of acceptance.
  Change= (One week after the intervention score - Baseline score)
Change from baseline in the score of acceptance assessed by Acceptance and Action Cancer Questionnaire at three months after the intervention | Baseline (T0) and three months follow-up (T2, three months after the 4-week intervention)
  18-item questionnaire to measure experiential avoidance, in which participants response the possibility that they accept or avoid repulsive thoughts and feelings to each item using a 7-point Likert scale (1 = never true to 7 = always true) ranged from 18 to 126. The higher the overall score, the greater level of experiential avoidance or low level of acceptance. 18 indicates low level of acceptance and 90 indicates the high level of acceptance.
  Change= (Three months after the intervention score - Baseline score)
Change from baseline in the score of cognitive fusion assessed by Cognitive Fusion Questionnaire at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 4-week intervention)
  An instrument to measure cognitive fusion, one of the components in the model of psychopathology of ACT. It has 9 items scored by 7-point Liker scale (1 = never true to 7 = always true) ranged from 9 to 63. 9 indicates low level of cognitive fusion and 63 indicates the high level of cognitive fusion.
  Change= (One week after the intervention score - Baseline score)
Change from baseline in the score of cognitive fusion assessed by Cognitive Fusion Questionnaire at three months after the intervention | Baseline (T0) and three months follow-up (T2, three months after the 4-week intervention)
  An instrument to measure cognitive fusion, one of the components in the model of psychopathology of ACT. It has 9 items scored by 7-point Liker scale (1 = never true to 7 = always true) ranged from 9 to 63. 9 indicates low level of cognitive fusion and 63 indicates the high level of cognitive fusion.
  Change= (Three months after the intervention score - Baseline score)

CONTACTS AND LOCATIONS:
Overall Officials: Huiyuan LI, Principal Investigator — Chinese University of Hong Kong; Cho Lee Wong, PhD, Study Director — Chinese University of Hong Kong
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No